CLINICAL TRIAL: NCT04427735
Title: Effect of Covid-19 Epidemic on Primary PCI and Prognosis in Patients With Acute STEMI
Brief Title: Effect of Covid-19 Epidemic on Primary PCI in Patients With STEMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hongwei Li, MD, professor, Beijing Friendship Hospital
Other Study IDs: BFH-COVID-19 and Primary PCI
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: STEMI
Keywords: covid-19; STEMI; primary PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; COVID-19

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- before COVID-19: Patients with myocardial infarction from January 24, 2019 to June 24, 2019
- after COVID-19: Patients with myocardial infarction from January 24, 2020 to June 24, 2020

SUMMARY:
The epidemic of covid-19 has spread all over the world and has a great impact on people's health and life. It is necessary to study the treatment of STEMI patients in the real world under the influence of the epidemic,which provide effective suggestions and strategies for emergency and severe treatment.

DETAILED DESCRIPTION:
The epidemic of covid-19 has spread all over the world and has a great impact on people's health and life. The patients' prognosis is poor because the epidemic situation runs on medical resources, delays the diagnosis and treatment of other diseases such as cardiovascular diseases, and the patients' willingness to see a doctor is reduced. In particular, the delay in the treatment of STEMI, which needs PCI treatment, will cause more damage to the patients. It is necessary to study the treatment of STEMI patients in the real world under the influence of the epidemic. In this study, STEMI patients who experienced emergency PCI treatment after the covid-19 outbreak in 2020 were included, and compared with the data of the same period in 2019,we will analyze the pre hospital treatment time, vascular opening time,and the major cardiovascular adverse events, which provide effective suggestions and strategies for emergency and severe treatment.

ELIGIBILITY:
Inclusion Criteria:

* Continuous inclusion of patients with definite diagnosis of acute ST segment elevation myocardial infarction and emergency PCI intervention.

Exclusion Criteria:

* Febrile patients, patients with severe infection,
* ST segment elevation myocardial infarction during hospitalization,
* Patients who could not cooperate with each other.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with definite diagnosis of acute ST segment elevation myocardial infarction and emergency PCI intervention
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-07-24 (Estimated); Study Completion 2021-07-24 (Estimated)

PRIMARY OUTCOMES:
MACE (major adverse cardiovascular events) | 1 year
  cardiovascular death, re-infarction, malignant arrhythmia,heart failure, revascularization, and stroke
all-cause death | 1 year
  death caused by all reason

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Li, Study Chair — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Gong X, Zhou L, Dong T, Ding X, Zhao H, Chen H, Li H. Impact of COVID-19 pandemic on STEMI undergoing primary PCI treatment in Beijing, China. Am J Emerg Med. 2022 Mar;53:68-72. doi: 10.1016/j.ajem.2021.11.034. Epub 2021 Nov 24. PMID 34999563